CLINICAL TRIAL: NCT01321333
Title: A Phase I/II Study of the Safety and Preliminary Efficacy of Intramedullary Spinal Cord Transplantation of Human Central Nervous System (CNS) Stem Cells (HuCNS-SC®) in Subjects With Thoracic (T2-T11) Spinal Cord Trauma
Brief Title: Study of Human Central Nervous System Stem Cells (HuCNS-SC) in Patients With Thoracic Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-N02-SC
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Thoracic Spinal Cord Injury; Spinal Cord Injury; Spinal Cord Injury Thoracic; Spinal Cord Trauma
Keywords: thoracic spinal cord injury; spinal cord injury thoracic; sub-acute spinal cord injury; human neural stem cells; stem cells; stem cells transplant; stem cells transplant spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC cells (Experimental): Single dose intramedullary administration of HuCNS-SC cells
  Interventions: Biological: HuCNS-SC cells

INTERVENTIONS:
Biological: HuCNS-SC cells — single dose intramedullary transplantation of HuCNS-SC cells in the thoracic spinal cord
  Other Names: Human central nervous system stem cells; allogeneic stem cells

SUMMARY:
This study will evaluate the effect of single transplantation of HuCNS-SC cells into the thoracic spinal cord of patients with sub-acute spinal cord injury.

DETAILED DESCRIPTION:
Study subjects will receive immunosuppression for nine months following transplantation. All enrolled subjects will be followed for one year following transplantation and then will be enrolled in a separate long-term follow-up study for an additional four years.

ELIGIBILITY:
Inclusion Criteria:

* T2-T11 thoracic spinal cord injury based on American Spinal Injury Association (ASIA) level determination by the principal investigator (PI)
* T2-T11 thoracic spinal cord injury as assessed by magnetic resonance imaging (MRI) and/or computerized tomography (CT)
* ASIA Impairment Scale (AIS) Grade A, B, or C
* Minimum of six weeks post injury for the initiation of screening
* Must have evidence of preserved conus function
* Must be at stable stage of medical recovery after injury

Exclusion Criteria:

* History of traumatic brain injury without recovery
* Penetrating spinal cord injury
* Evidence of spinal instability or persistent spinal stenosis and/or compression related to initial trauma
* Previous organ, tissue or bone marrow transplantation
* Previous participation in any gene transfer or cell transplant trial
* Current or prior malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Types and frequencies of adverse events and serious adverse events | One year after transplant
  Analysis of types and frequencies of adverse events one year after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Chair — StemCells, Inc.
Locations (3):
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - Toronto Western Hospital, Toronto, Ontario
- University Hospital Balgrist- Uniklinik Balgrist, Forschstrasse 340, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: Click here for more information on this study — http://www.stemcellsinc.com/Therapeutic-Programs/Overview.htm